CLINICAL TRIAL: NCT00946933
Title: Effects of Chronic Acid-Base Changes on the Ventilatory and Perceptual Response to Hypercapnia, Hypoxia and Exercise in Healthy Older Adults
Brief Title: Effects of Chronic Acid-Base Changes on Ventilatory and Perceptual Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DSS-16198
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: acid-base balance; ventilatory control; dyspnea; exercise; modified rebreathing procedure; Normal; older
MeSH Terms: conditions — Dyspnea; Motor Activity | interventions — Ammonium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 0.025 g/kg/day of NaCl (sodium chloride)
  Interventions: Dietary Supplement: placebo
- High salt diet (Active Comparator): 0.2 g/kg/day of NH4Cl (ammonium chloride)
  Interventions: Dietary Supplement: NH4Cl (ammonium chloride)

INTERVENTIONS:
Dietary Supplement: NH4Cl (ammonium chloride) — 0.2 g/kg/day of NH4Cl (ammonium chloride)
  Arms: High salt diet
Dietary Supplement: placebo — 0.025 g/kg/day of NaCl (sodium chloride)
  Arms: Placebo

SUMMARY:
Approximately 30% of people aged 65 years and older experience breathlessness (perceived respiratory difficulty) during daily activity. The main causes of increased breathlessness in the healthy elderly are poorly understood and are the main focus of the proposed study. Some possible contributing factors include abnormalities in the control and/or mechanics of breathing. To evaluate these possible contributory factors, the investigators will compare ventilatory and perceptual responses to: 1) exercise, 2) increased levels of inspired carbon dioxide, and 3) reduced levels of inspired oxygen under strictly-controlled experimental conditions where the investigators increase or decrease breathing requirements by altering dietary salt intake in healthy 40-80 year old men and women.

Exercise and rebreathing tests will be performed at baseline and at the end of each 3 day treatment period. Breathlessness intensity will be measured and compared at a standardized work rate, ventilation or end-tidal PCO2 during these tests.

ELIGIBILITY:
Inclusion Criteria:

* healthy, regularly active adults
* non-smoking
* BMI 18-30 kg/m2

Exclusion Criteria:

* history of lung and/or heart disease (including cardiac arrhythmias) or other comorbidity which could interfere with proper conduct of the intervention or tests
* hypotension or hypertension
* hypercholesterolemia
* sleep disordered breathing
* inability to perform cycle exercise or comply with other testing procedures

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Breathlessness intensity (10-point Borg scale) | Measured at the end of each 3 day treatment period

SECONDARY OUTCOMES:
Exercise capacity (peak VO2) | Measured at the end of each 3 day treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Respiratory Investigation Unit at Kingston General Hospital, Kingston, Ontario, Canada